CLINICAL TRIAL: NCT02358538
Title: A Multicenter, Open-Label Proof-of-Concept Trial of Ganaxolone in Children With PCDH19 Female Pediatric Epilepsy and Other Rare Genetic Epilepsies Followed by 52 Week Open-Label Treatment
Brief Title: Open-Label PoC Trial of Ganaxolone in Children With PCDH19 Female Pediatric Epilepsy and Other Rare Genetic Epilepsies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1042-900
Record Dates: First submitted 2015-01-30; First posted 2015-02-09 (Estimated); Results first posted 2022-09-07 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Epilepsy
Keywords: PCDH19; ganaxolone; neurosteroid; CDKL5; LGS; CSWS
MeSH Terms: conditions — Epilepsy | interventions — ganaxolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ganaxolone (Experimental): Maximum of 1800 mg/day or 63 mg/kg/day
  Interventions: Drug: Ganaxolone

INTERVENTIONS:
Drug: Ganaxolone — oral suspension or capsules
  Other Names: CCD 1042

SUMMARY:
To evaluate the efficacy of open-label ganaxolone as adjunctive therapy for uncontrolled seizures in female children with PCDH19 mutation and other rare genetic epilepsies in an open-label proof-of-concept study.

DETAILED DESCRIPTION:
The purpose of this proof-of-concept study is to evaluate ganaxolone as adjunctive therapy for uncontrolled seizures in female children with PCDH19 mutations and other rare genetic epilepsies. After establishing baseline seizure frequency, qualifying subjects will enter the study and be treated with open-label ganaxolone for up to six months.

ELIGIBILITY:
Key Inclusion Criteria:

1. Have parent or legal guardian available and willing to give written informed consent.
2. Male and female outpatients between 2 and 18 years of age years of age at time of consent.
3. Have any of the following epilepsy syndromes: PCDH19; CDKL5; Dravet Syndrome; Lennox Gastaut Syndrome (LGS); Continuous Spikes and Waves during Sleep (CSWS)
4. Have uncontrolled cluster seizures and/or non-clustered seizures.
5. Subjects should be on a stable regimen of anti-epileptic medication, and generally in good health.
6. Parent or guardian is able and willing to maintain an accurate and complete daily written seizure calendar.
7. Able and willing to take study medication with food, two or three times daily.

Key Exclusion Criteria

1. Have had previous exposure to ganaxolone.
2. Known sensitivity or allergy to any component in the study drug, progesterone, or other related steroid compounds.
3. Exposure to any investigational drug or device < 90 days prior to screening, or plans to participate in another drug or device trial at any time during the study.
4. Concurrent use of vigabatrin, tiagabine, or ezogabine is not permitted.
5. Have any medical condition that, in the investigator's judgment, is considered to be clinically significant and could potentially affect subject safety or study outcome, including but not limited to: clinically significant cardiac, renal, pulmonary, gastrointestinal, hematologic or hepatic conditions; or a condition that affects the absorption, distribution, metabolism or excretion of drugs.
6. Have active suicidal plan/intent, or have had active suicidal thoughts in the past 6 months or a suicide attempt in the past 3 years.
7. Have Alanine transferase (ALT; SGPT) or Aspartate transferase (AST; SGOT) levels > 3 times upper limits of normal (ULN), or total bilirubin >1.5 time ULN at the screening and baseline visits.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2019-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Sutter Institute for Medical Research, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Center for Rare Neurological Diseases, Norcross, Georgia
  - JWM Neurology, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Institute of Neurology and Neurosurgery at St. Barnabas, Livingston, New Jersey
  - Nationwide Children's Hospital, Columbus, Ohio
- Bambino Gesu Children's Hospital, IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period May 08, 2015
Groups:
- CDKL5: Cyclin-dependent kinase-like 5
- CSWS: Continuous Spike Wave in Sleep
- Lennox-Gastaut: Lennox-Gastaut Syndrome pediatric epilepsy
- PCDH19: Protocadherin-19
Period: Through Week 26
Arm/Group | CDKL5 | CSWS | Lennox-Gastaut | PCDH19
Started | 7 | 2 | 10 | 11
Completed | 4 | 0 | 5 | 6
Not Completed | 3 | 2 | 5 | 5
Not completed — Adverse Event | 0 | 1 | 1 | 2
Not completed — Lack of Efficacy | 1 | 1 | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Non-Compliance | 0 | 0 | 1 | 0
Not completed — Family did not see benefit from IP | 1 | 0 | 0 | 0
Period: 52 Week Extension Period
Arm/Group | CDKL5 | CSWS | Lennox-Gastaut | PCDH19
Started | 4 | 0 | 4 | 6
Completed | 4 | 0 | 2 | 2
Not Completed | 0 | 0 | 2 | 4
Not completed — Lack of Efficacy | 0 | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Population: MITT population
Groups:
- CSWS: Continuous Spike and Waves during Sleep
- Lennox- Gastaut: Lennox- Gastaut syndrome
- Total: Total of all reporting groups
Arm/Group | CDKL5 | CSWS | Lennox- Gastaut | PCDH19 | Total
Number analyzed (Participants) | 7 | 2 | 10 | 11 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 2 | 10 | 11 | 30
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.57 (5.167) | 11.55 (5.728) | 9.12 (2.352) | 9.00 (3.956) | 8.88 (3.834)
Age, Continuous [Mean (Standard Deviation); unit: years] — Age - Safety population in the 52-week open label extension period Population: Content is associated with 52-week open label period (as the label indicates)
  years
    number analyzed (Participants) | 4 | 0 | 4 | 6 | 14
    (all) | 7.73 (3.403) |  | 9.25 (3.595) | 8.87 (4.129) | 8.65 (3.551)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7 | 11 | 25
  Male | 1 | 1 | 3 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants] — Gender - Safety population in the 52-week open label extension period Population: Content is associated with 52-week open label period (as the label indicates)
  Participants
    number analyzed (Participants) | 4 | 0 | 4 | 6 | 14
    Female | 4 |  | 4 | 6 | 14
    Male | 0 |  | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 4 | 3 | 7
  Not Hispanic or Latino | 7 | 2 | 6 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity - Safety population in the 52-week open label extension period Population: Content is associated with 52-week open label period (as the label indicates)
  Participants
    number analyzed (Participants) | 4 | 0 | 4 | 6 | 14
    Hispanic or Latino | 0 |  | 2 | 2 | 4
    Not Hispanic or Latino | 4 |  | 2 | 4 | 10
    Unknown or Not Reported | 0 |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 7 | 1 | 4 | 10 | 22
  More than one race | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race - Safety population in the 52-week open label extension period Population: Content is associated with 52-week open label period (as the label indicates)
  Participants
    number analyzed (Participants) | 4 | 0 | 4 | 6 | 14
    American Indian or Alaska Native | 0 |  | 0 | 0 | 0
    Asian | 0 |  | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0 | 0
    Black or African American | 0 |  | 1 | 0 | 1
    White | 4 |  | 1 | 6 | 11
    More than one race | 0 |  | 2 | 0 | 2
    Unknown or Not Reported | 0 |  | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Summary of 28-day Seizure Frequency for Sum of Individual Seizures and Clusters for 52-week OLE Period (Mean Percent Change & Standard Deviation)
Description: Percentage change from baseline in 28-day seizure frequency at 3 months (day 91), 26 weeks, 52 week OLE (Mean Percent Change & Standard Deviation)
Time Frame: Baseline through 52 week open label period
Population: MITT Population
Measure: Mean (Standard Deviation); unit: percentage of change of frequency
Arm/Group | CDKL5 | CSWS | Lennox- Gastaut | PCDH19
Number analyzed (Participants) | 7 | 2 | 10 | 11
percentage of change of frequency
  Percent Change from baseline (at day 91) | -31.23 (41.438) | NA (NA) — Both patients (2 for CSWS) discontinued so data is not available. | 122.10 (321.124) | 52.83 (234.084)
  Percent Change from baseline (at week 26) | -20.55 (60.588) | NA (NA) — Both patients (2 for CSWS) discontinued so data is not available. | 125.38 (319.051) | 46.36 (235.661)
  Percent change from baseline (52 week OLE through month 6): number analyzed (Participants) | 4 | 2 | 2 | 6
  Percent change from baseline (52 week OLE through month 6) | -54.41 (40.286) | NA (NA) — Both patients (2 for CSWS) discontinued so data is not available. | -38.74 (9.292) | -19.98 (63.644)
  Percent change from baseline (52 week OLE period): number analyzed (Participants) | 4 | 2 | 2 | 6
  Percent change from baseline (52 week OLE period) | -49.20 (50.206) | NA (NA) — Both patients (2 for CSWS) discontinued so data is not available. | -37.75 (7.891) | -19.95 (63.571)

2. Primary Outcome: Summary of 28-day Seizure Frequency for Sum of Individual Seizures and Clusters Through 52-week OLE (Median Percent Change)
Description: Percentage change from baseline in 28-day seizure frequency at 3 months (day 91), 26 weeks, 52 week OLE (Median Percent Change)
Time Frame: Baseline through 52-week open- label period
Population: MITT Population
Measure: Median (Full Range); unit: Median Percent Change in Frequency
Arm/Group | CDKL5 | Lennox-Gastaut | PCDH19 | CSWS
Number analyzed (Participants) | 7 | 10 | 11 | 2
Median Percent Change in Frequency
  Percent change from baseline (at Day 91) | -47.34 [-80.9 to 36.8] | -10.22 [-68.1 to 904.3] | -25.98 [-100.00 to 723.2] | NA [NA to NA] — Both patients (2 for CSWS) discontinued so data is not available.
  Percent change from baseline (at week 26) | -37.70 [-85.3 to 99.9] | -9.19 [-71.2 to 904.3] | -24.59 [-100.00 to 723.2] | NA [NA to NA] — Both patients (2 for CSWS) discontinued so data is not available.
  Percent change from baseline (at week 26) - with 6 duplicate diary entries removed | -44.4 [-85.3 to 99.9] | NA [NA to NA] — There is no data available to support this row for this ARM. One subject in the CDKL5 cohort had duplications of data on 6 days. These data appeared to the investigator and sponsor to be erroneous. Excluding these days changes the median percent change from baseline at Week 26 to 44.4 for the CDKL5 cohort. This is reflected in the CDKL5 ARM. | NA [NA to NA] — There is no data available to support this row for this ARM. One subject in the CDKL5 cohort had duplications of data on 6 days. These data appeared to the investigator and sponsor to be erroneous. Excluding these days changes the median percent change from baseline at Week 26 to 44.4 for the CDKL5 cohort. This is reflected in the CDKL5 ARM. | NA [NA to NA] — Both patients (2 for CSWS) discontinued so data is not available.
  Percent change from baseline (52 week OLE through month 6): number analyzed (Participants) | 4 | 10 | 2 | 2
  Percent change from baseline (52 week OLE through month 6) | -58.94 [-89.4 to -10.4] | -38.74 [-45.3 to -32.2] | -13.48 [-100.0 to 59.6] | NA [NA to NA] — Both patients (2 for CSWS) discontinued so data is not available.
  Percent change from baseline (52 week OLE period) | -61.93 [-89.5 to 16.6] | -37.75 [-43.3 to -32.2] | -13.48 [-99.0 to 59.6] | NA [NA to NA] — Both patients (2 for CSWS) discontinued so data is not available.

3. Secondary Outcome: Summary of CGII-C
Description: Clinician Global Impression of Change score as assessed by questionnaire. [ Time Frame: 78 Weeks ] CGII-C scale is qualitative values and not quantitative.
Time Frame: End of Week 4, End of Week 8, End of Week 17, End of Week 26, Week 44, Week 62, Week 78
Population: MITT Population - n varies per visit, also CSWS is not included
Measure: Count of Participants; unit: Participants
Arm/Group | CDKL5 | Lennox-Gastaut | PCDH19 | CSWS
Number analyzed (Participants) | 7 | 10 | 11 | 2
Participants
  Visit 4 (End of Week 4) - Very Much Improved: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - Very Much Improved | 0 | 2 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 4 (End of Week 4) - Much Improved: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - Much Improved | 3 | 4 | 4 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 4 (End of Week 4) - Minimally Improved: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - Minimally Improved | 2 | 2 | 3 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 4 (End of Week 4) - No Change: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - No Change | 2 | 0 | 3 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 4 (End of Week 4) - Minimally Worse: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - Minimally Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 4 (End of Week 4) - Much Worse: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 4 (End of Week 4) - Very Much Worse: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - Very Much Improved: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - Very Much Improved | 0 | 1 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - Much Improved: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - Much Improved | 4 | 4 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - Minimally Improved: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - Minimally Improved | 2 | 2 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - No Change: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - No Change | 1 | 1 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - Minimally Worse: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - Minimally Worse | 0 | 0 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - Much Worse: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - Very Much Worse: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - Very Much Improved: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - Very Much Improved | 1 | 2 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - Much Improved: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - Much Improved | 2 | 3 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - Minimally Improved: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - Minimally Improved | 2 | 0 | 4 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - No Change: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - No Change | 0 | 1 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - Minimally Worse: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - Minimally Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - Much Worse: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - Very Much Worse: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - Very Much Improved: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - Very Much Improved | 0 | 1 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - Much Improved: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - Much Improved | 3 | 1 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - Minimally Improved: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - Minimally Improved | 1 | 1 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - No Change: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - No Change | 2 | 2 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - Minimally Worse: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - Minimally Worse | 0 | 1 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - Much Worse: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - Much Worse | 1 | 1 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - Very Much Worse: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - Very Much Improved: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - Very Much Improved | 0 | 0 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - Much Improved: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - Much Improved | 3 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - Minimally Improved: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - Minimally Improved | 1 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - No Change: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - No Change | 0 | 1 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - Minimally Worse: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - Minimally Worse | 0 | 1 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - Much Worse: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - Very Much Worse: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - Very Much Improved: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - Very Much Improved | 0 | 0 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - Much Improved: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - Much Improved | 4 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - Minimally Improved: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - Minimally Improved | 0 | 1 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - No Change: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - No Change | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - Minimally Worse: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - Minimally Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - Much Worse: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - Very Much Worse: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - Very Much Improved: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - Very Much Improved | 0 | 0 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - Much Improved: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - Much Improved | 3 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - Minimally Improved: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - Minimally Improved | 0 | 1 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - No Change: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - No Change | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - Minimally Worse: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - Minimally Worse | 0 | 0 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - Much Worse: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - Much Worse | 0 | 0 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - Very Much Worse: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.

4. Secondary Outcome: Summary of CGII-P
Description: Patient Global Impression of Change score as assessed by questionnaire. [ Time Frame: 78 Weeks ] CGII-P scale is qualitative values and not quantitative.
Time Frame: Patient Global Impression of Change score as assessed by questionnaire. [ Time Frame: 78 Weeks ]
Population: MITT Population - n varies per visit, also CSWS is not included
Measure: Count of Participants; unit: Participants
Arm/Group | CDKL5 | Lennox-Gastaut | PCDH19 | CSWS
Number analyzed (Participants) | 7 | 10 | 11 | 2
Participants
  Visit 4 (End of Week 4) - Very Much Improved: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - Very Much Improved | 0 | 3 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 4 (End of Week 4) - Much Improved: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - Much Improved | 1 | 2 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 4 (End of Week 4) - Minimally Improved: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - Minimally Improved | 4 | 3 | 5 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 4 (End of Week 4) - No Change: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - No Change | 2 | 0 | 3 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 4 (End of Week 4) - Minimally Worse: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - Minimally Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 4 (End of Week 4) - Much Worse: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 4 (End of Week 4) - Very Much Worse: number analyzed (Participants) | 7 | 8 | 11 | 2
  Visit 4 (End of Week 4) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - Very Much Improved: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - Very Much Improved | 0 | 2 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - Much Improved: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - Much Improved | 1 | 2 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - Minimally Improved: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - Minimally Improved | 5 | 3 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - No Change: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - No Change | 0 | 1 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - Minimally Worse: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - Minimally Worse | 1 | 0 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - Much Worse: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - Much Worse | 0 | 0 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 5 (End of Week 8) - Very Much Worse: number analyzed (Participants) | 7 | 8 | 7 | 2
  Visit 5 (End of Week 8) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - Very Much Improved: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - Very Much Improved | 1 | 1 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - Much Improved: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - Much Improved | 2 | 1 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - Minimally Improved: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - Minimally Improved | 2 | 3 | 4 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - No Change: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - No Change | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - Minimally Worse: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - Minimally Worse | 0 | 1 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - Much Worse: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 6 (End of Week 17) - Very Much Worse: number analyzed (Participants) | 5 | 6 | 6 | 2
  Visit 6 (End of Week 17) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - Very Much Improved: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - Very Much Improved | 0 | 1 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - Much Improved: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - Much Improved | 4 | 1 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - Minimally Improved: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - Minimally Improved | 0 | 3 | 3 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - No Change: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - No Change | 1 | 1 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - Minimally Worse: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - Minimally Worse | 1 | 0 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - Much Worse: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - Much Worse | 1 | 1 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 7 (End of Week 26) - Very Much Worse: number analyzed (Participants) | 7 | 7 | 9 | 2
  Visit 7 (End of Week 26) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - Very Much Improved: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - Very Much Improved | 0 | 0 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - Much Improved: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - Much Improved | 2 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - Minimally Improved: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - Minimally Improved | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - No Change: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - No Change | 2 | 1 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - Minimally Worse: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - Minimally Worse | 0 | 1 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44) - Much Worse: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44) - Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 8 (End of Week 44)- Very Much Worse: number analyzed (Participants) | 4 | 2 | 2 | 2
  Visit 8 (End of Week 44)- Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - Very Much Improved: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - Very Much Improved | 2 | 0 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - Much Improved: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - Much Improved | 2 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62)- Minimally Improved: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62)- Minimally Improved | 0 | 1 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - No Change: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - No Change | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - Minimally Worse: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - Minimally Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - Much Worse: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 9 (End of Week 62) - Very Much Worse: number analyzed (Participants) | 4 | 1 | 2 | 2
  Visit 9 (End of Week 62) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - Very Much Improved: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - Very Much Improved | 1 | 0 | 2 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - Much Improved: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - Much Improved | 2 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78)- Minimally Improved: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78)- Minimally Improved | 0 | 1 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - No Change: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - No Change | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - Minimally Worse: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - Minimally Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - Much Worse: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - Much Worse | 0 | 0 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Visit 10 (End of Week 78) - Very Much Worse: number analyzed (Participants) | 3 | 1 | 4 | 2
  Visit 10 (End of Week 78) - Very Much Worse | 0 | 0 | 0 | NA — Both patients (2 for CSWS) discontinued so data is not available.

5. Secondary Outcome: Number of Participants With Responder Rate of Seizure Frequency
Description: Responder Rate in Terms of 28-day Seizure Frequency Based on the Sum of Individual Seizures and Clusters
Time Frame: Month 3 and Week 26
Population: MITT Population - n varies per visit, also CSWS is not included
Measure: Count of Participants; unit: Participants
Arm/Group | CDKL5 | Lennox-Gastaut | PCDH19 | CSWS
Number analyzed (Participants) | 7 | 10 | 11 | 2
Participants
  Post-baseline through Month 3 (Day 91) - 25% Responder | 4 | 4 | 6 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Post-baseline through Month 3 (Day 91) - 50% Responder | 3 | 2 | 4 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Post-baseline through Month 3 (Day 91) - 75% Responder | 1 | 0 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Post-baseline 26-week open-label Period - 25% Responder | 4 | 3 | 5 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Post-baseline 26-week open-label Period - 50% Responder | 2 | 1 | 3 | NA — Both patients (2 for CSWS) discontinued so data is not available.
  Post-baseline 26-week open-label Period - 75% Responder | 1 | 0 | 1 | NA — Both patients (2 for CSWS) discontinued so data is not available.

6. Secondary Outcome: Mean Percentage Change of Individual Seizure-free Days
Description: Mean Percentage Change of Individual Seizure-free days per 28-day period (through 52-week OLE) period relative to baseline
Time Frame: Baseline, Day 91, Week 26, 52-week OLE through month 6, 52-week OLE Period
Population: MITT Population - n varies per visit, also CSWS is not included
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | CDKL5 | Lennox-Gastaut | PCDH19 | CSWS
Number analyzed (Participants) | 7 | 10 | 11 | 2
Percentage Change
  Mean Percentage Change of individual seizure-free days from baseline to Day 91 | 11.84 (18.472) | -1.12 (24.928) | 7.87 (17.843) | NA (NA) — Both patients (2 for CSWS) discontinued so data is not available.
  Mean Percentage Change of individual seizure-free days from baseline to Week 26 | 11.80 (20.968) | -2.13 (22.042) | 7.94 (18.016) | NA (NA) — Both patients (2 for CSWS) discontinued so data is not available.
  Mean Percentage Change of individual seizure-free days from baseline to 52-week OLE (181 days): number analyzed (Participants) | 4 | 2 | 6 | 2
  Mean Percentage Change of individual seizure-free days from baseline to 52-week OLE (181 days) | 21 (30.85) | 16.35 (2.916) | 17.12 (27.040) | NA (NA) — Both patients (2 for CSWS) discontinued so data is not available.
  Mean Percentage Change of individual seizure-free days from baseline to 52-week OLE Period: number analyzed (Participants) | 4 | 2 | 6 | 2
  Mean Percentage Change of individual seizure-free days from baseline to 52-week OLE Period | 20.44 (28.788) | 14.95 (4.897) | 17.02 (26.904) | NA (NA) — Both patients (2 for CSWS) discontinued so data is not available.

ADVERSE EVENTS:
Time Frame: Combined 26-week open label period and 52-week open label extension period
Description: Overall Summary of Adverse Events (Safety Population)
Arm/Group | CDKL5 | CSWS | Lennox-Gastaut | PCDH19
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/2 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/2 | 2/10 | 3/11
Other Adverse Events (participants affected / at risk) | 7/7 | 1/2 | 7/10 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDKL5 (N=7) | CSWS (N=2) | Lennox-Gastaut (N=10) | PCDH19 (N=11)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Unintentional Medical Device Removal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDKL5 (N=7) | CSWS (N=2) | Lennox-Gastaut (N=10) | PCDH19 (N=11)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 2 (4) | 4 (6)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 5 (22) | 0 (0) | 1 (2) | 7 (16)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (8) | 0 (0) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 2 (5) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (9) | 1 (1) | 1 (3) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abnormal behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Balance Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fungal Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Enuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrostomy (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
CSWS cohort was not included in efficacy summaries as only 2 subjects were enrolled in cohort; however, cohort was included in the subject data listings.

Overall number of participants affected is associated with all TEAEs and not >-5%. Individual AEs are associated with >-5%.

One patient in the CDKL5 cohort had duplication of data on 6 days, which appeared to PI and sponsor to be erroneous. This datapoint is represented accordingly in outcome measure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT02358538/Prot_002.pdf
  • Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT02358538/SAP_003.pdf